CLINICAL TRIAL: NCT00036517
Title: A Phase I/IIA, Multicenter, Double-Blind, Randomized, Placebo-Controlled, Crossover, Dose Escalation, Safety Study of the Chemotherapy Modulator PHY906 in Patients With Advanced Colorectal Cancer
Brief Title: Safety Study of the Chemotherapy Modulator PHY906 in Patients With Advanced Colorectal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PhytoCeutica (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PHY906-2000-1
Record Dates: First submitted 2002-05-10; First posted 2002-05-13 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-09

CONDITIONS: Colorectal Neoplasms; Diarrhea
Keywords: Stage III and Stage IV colorectal cancer; diarrhea; reduce; alleviate; modulate; Saltz regimen; CPT-11; irinotecan; camptosar; 5-fluorouracil; leucovorin; 5-FU; LV; chemotherapy; side effect; toxicity; botanical drug; herbal medicine; chinese herbal medicine; traditional chinese medicine; TCM; oral dose; oral administration; concomitant use
MeSH Terms: conditions — Colorectal Neoplasms; Diarrhea | interventions — PHY 906

INTERVENTIONS:
Drug: PHY906

SUMMARY:
The triple combination chemotherapy of irinotecan, 5-fluorouracil and leucovorin (CPT-11/5-FU/LV or Saltz regimen) is the treatment of choice for patients with advanced colorectal cancer. Severe diarrhea, unfortunately, is a side effect of such treatment. Preclinical studies have indicated that the botanical drug PHY906 can reduce such diarrhea without compromising the effectiveness of the chemotherapy. The primary purpose of this clinical study is to evaluate the safety, tolerability and minimum effective dose of PHY906 when administered in conjunction with the Saltz regimen.

DETAILED DESCRIPTION:
CPT-11/5-FU/LV is an active combination agent in the treatment of colorectal cancer, but one of its dose-limiting toxicities is diarrhea. PHY906 has been shown to reduce the severity of CPT-11-induced toxicity without compromising antitumor efficacy in in vivo animal models. Additionally, there has been a long historical experience in the Far East demonstrating safety of PHY906 in humans. Thus, we are conducting this double-blind, placebo-controlled study to evaluate the safety and tolerability of PHY906. This dose escalation study will also examine the effect of PHY906 (1.2, 2.4, and 3.6 g/day) on the pharmacokinetics of CPT-11 and 5-FU after concomitant administration with CPT-11, 5-FU, and LV, and on the severity of CPT-11-induced toxicities such as diarrhea.

ELIGIBILITY:
Inclusion Criteria

Patients must:

* be between 18 and 75 years of age, inclusive, at the time of enrollment.
* have advanced colorectal carcinoma, which may be either measurable or non-measurable.
* not have received either CPT-11, FU, or other cytotoxic chemotherapy agents in any setting (including adjuvant) within 1 year prior to screening.
* have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* use an effective contraceptive method if the patients are of reproductive potential while enrolled in the study, since the potential effects of the herbs on a developing fetus are unknown.
* have an estimated life expectancy of at least 20 weeks.
* provide written informed consent.
* have adequate organ function as indicated by the following laboratory values; these laboratory values must be obtained within 14 days prior to study enrollment:
* Bone marrow reserve: absolute granulocyte count (AGC) more than or equal to 1.5 X 10(to the power of 9)/L, platelet count more than or equal to 100 X 10 (to the power of 9)/L, and hemoglobin level more than or equal to 9 g/dL.
* Hepatic function: serum total bilirubin concentration no greater than 1.5 mg/dL, aspartate transaminase (AST or serum glutamic-oxaloacetic transaminase [SGOT]), and alanine transaminase (ALT or serum glutamic-pyruvic transaminase [SGPT]) levels no greater than grade 2 toxicity as determined from the NCI-CTC version 2.0.
* Renal function: serum creatinine level no greater than grade 2 toxicity as determined from the CTC version 2.0.

Exclusion Criteria

Patients who have or are:

* Gilbert syndrome (familial, non-hemolytic, acholuric jaundice).
* patients with enterostomies.
* untreated brain metastases or deteriorating neurological function after the completion of cranial irradiation.
* a woman who is currently pregnant and/or breast-feeding.
* active infections or any serious systemic disorder that, in the opinion of the principal investigator, are incompatible with the study product and/or procedures.
* used an investigational agent within 4 weeks of study entry.
* a known hypersensitivity to the study medication, its excipients, its analogs, or any of the component herbs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2002-02; Study Completion 2003-03

CONTACTS AND LOCATIONS:
Overall Officials: Wayne D Brenckman, Jr., MD, Study Director — Inveresk Research
Locations (3):
- United States (3):
  - VA CT Cancer Center, West Haven, Connecticut
  - Weill Cornell Medical Center, New York, New York
  - Cancer Centers of the Carolinas, Greenville, South Carolina